CLINICAL TRIAL: NCT06700018
Title: Development of a Novel Method for Detailed Evaluation of Blood Flow Patterns in Stented Segments and Assessment of Their Role in Stent Thrombosis
Brief Title: Flow Patterns and Stent Thrombosis
Acronym: TISIS registry
Status: Recruiting | Type: Observational
Sponsor: Queen Mary University of London (Other)
Collaborators: Barts Helth NHS Trust (Unknown); Oxford University Hospitals NHS Trust (Other); Royal Free Hospital NHS Foundation Trust (Other); University Hospitals Bristol and Weston NHS Foundation Trust (Other); Mid and South Essex NHS Foundation Trust (Other); Newcastle-upon-Tyne Hospitals NHS Trust (Other); Liverpool Heart and Chest Hospital NHS Foundation Trust (Other); Manchester University NHS Foundation Trust (Other Government); King's College Hospital NHS Trust (Other); San Giovanni Addolorata Hospital (Other); Medstar Health Research Institute (Other); Medical University of Warsaw (Other); Insel Gruppe AG, University Hospital Bern (Other); Hospital San Carlos, Madrid (Other); The Leeds Teaching Hospitals NHS Trust (Other); McMaster University Health Sciences Centre (Unknown); Fujita Health University (Other); Harbin Medical University (Other); Yale University (Other); Fundación de Investigación Biomédica - Hospital Universitario de La Princesa (Other); Erasmus Medical Center (Other); Radbound University Medical Center (Unknown); Department of Cardiovascular Surgery, German Heart Center Munich (Unknown); Columbia University (Other); The Queen Elizabeth Hospital (Other); Yonsei University Hospital, Seoul, South Korea (Unknown); Nara Medical University (Other); Shinshu University School of Medicine (Unknown); University Hospitals Sussex NHS Foundation Trust (Unknown); Galeazzi Sant'Ambrogio Hospital - Milan (Unknown); CORRIB Core Lab, University of Galway (Unknown)
Responsible Party: Sponsor
Other Study IDs: 331221
Record Dates: First submitted 2024-10-21; First posted 2024-11-21 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Stent Thrombosis
Keywords: stent thrombosis; endothelial shear stress; optical coherence tomography; blood flow simulations

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Stent thrombosis group: 40 patients who have suffered cardiovascular events attributed to stent thrombosis within one year of post-stent implementation will be recruited.
- Control group: 80 patients not having suffered stent thrombosis but will have uneventful follow-up. An effort will be made so that these patients have similar clinical presentation, baseline demographics and angiographic results post PCI and receive treatment with a similar antiplatelet regime compared to those who suffered stent thrombosis.

SUMMARY:
The goal of this observational study is to study the effect of haemodynamic forces on thrombus formation and identify haemodynamic markers that predict stent thrombosis events in patients who have undergone OCT-guided percutaneous coronary interventions.

The primary objective of the study is to examine the efficacy of blood flow patterns in predicting stent thrombosis. Researchers will compare the blood flow patterns of the stent thrombosis group with that of the control group to understand the influence of blood flow patterns on thrombus formation and progression.

DETAILED DESCRIPTION:
The incidences of Stent Thrombosis (ST) remain high in complex lesions and in high-risk patients. The use of intravascular imaging seems to be able to identify causes of ST, enabling prompt correction, and its use has been associated with better clinical outcomes in this setting. However, the efficacy of intravascular imaging features in predicting ST is limited. Computational fluid dynamic studies have shown that the local hemodynamic forces distribution has an effect on thrombus formation and can be responsible for the ST events. However, none of the studies today has explored in vivo the value of the flow disturbances in predicting events. The investigators have recently developed a method that is able to reconstruct vessel geometry accurately using coronary angiography and optical coherence tomography (OCT) data. Validation of this method in vitro and in human data showed promising results in accurately measuring shear stress and shear rate distribution.

This study, aims to explore the value of this method in predicting patients undergoing stent implantation with OCT imaging guidance that will suffer a ST. The investigators aim to collect data from 40 patients who had an ST after OCT-guided revascularization and from a control group of 80 patients who had no event after having stent implantation under OCT guidance. Investigators will further reconstruct the stented vessel from the OCT and the angiographic images, perform blood flow simulation and measure the shear rate and the shear stress in these two groups to explore the value of these metrics in predicting stent occlusion.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergone OCT-guided percutaneous coronary intervention and implanted with a second-generation drug-eluting stent
* Patients who have suffered thrombosis post-stent implantation

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: A total of 120 patients who have undergone OCT-guided percutaneous coronary intervention and implanted with a second-generation drug-eluting stent
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Haemodynamic shear stress and shear rate | 1.5 years
  The haemodynamic shear rate and shear rate will be calculated by performing CFD simulations on reconstructed geometries obtained from the percutaneous coronary interventions of the patients. The efficacy of the haemodynamic shear stress and shear rate in predicting stent thrombosis will be studied.

SECONDARY OUTCOMES:
OCT based stented segment reconstruction | 3 months
  To develop a methodology for the reconstruction of stented segments from OCT and angiographic data that relies on the separate modelling of the lumen and stent architecture and fusion of these geometries in a final model
Validation of the proposed reconstruction methodology | 4 months
  To validate in vivo and in-bench studies, the accuracy of the developed reconstruction method.
Development of automated frame work for reconstruction of stented segments | 6 months
  To design a user-friendly platform incorporating the new method to fast and accurately reconstruct vessels stented with different stent types.

CONTACTS AND LOCATIONS:
Locations (1):
- Queen Mary University of London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
The data sharing has not been decided yet. It may be considered in the future.

REFERENCES:
- [Background] Gijsen F, Katagiri Y, Barlis P, Bourantas C, Collet C, Coskun U, Daemen J, Dijkstra J, Edelman E, Evans P, van der Heiden K, Hose R, Koo BK, Krams R, Marsden A, Migliavacca F, Onuma Y, Ooi A, Poon E, Samady H, Stone P, Takahashi K, Tang D, Thondapu V, Tenekecioglu E, Timmins L, Torii R, Wentzel J, Serruys P. Expert recommendations on the assessment of wall shear stress in human coronary arteries: existing methodologies, technical considerations, and clinical applications. Eur Heart J. 2019 Nov 1;40(41):3421-3433. doi: 10.1093/eurheartj/ehz551. No abstract available. PMID 31566246
- [Background] Li Y, Li Z, Holck EN, Xu B, Karanasos A, Fei Z, Chang Y, Chu M, Dijkstra J, Christiansen EH, Reiber JHC, Holm NR, Tu S. Local Flow Patterns After Implantation of Bioresorbable Vascular Scaffold in Coronary Bifurcations - Novel Findings by Computational Fluid Dynamics. Circ J. 2018 May 25;82(6):1575-1583. doi: 10.1253/circj.CJ-17-1332. Epub 2018 Mar 24. PMID 29576586
- [Background] O'Brien CC, Kolandaivelu K, Brown J, Lopes AC, Kunio M, Kolachalama VB, Edelman ER. Constraining OCT with Knowledge of Device Design Enables High Accuracy Hemodynamic Assessment of Endovascular Implants. PLoS One. 2016 Feb 23;11(2):e0149178. doi: 10.1371/journal.pone.0149178. eCollection 2016. PMID 26906566
- [Background] Migliori S, Chiastra C, Bologna M, Montin E, Dubini G, Aurigemma C, Fedele R, Burzotta F, Mainardi L, Migliavacca F. A framework for computational fluid dynamic analyses of patient-specific stented coronary arteries from optical coherence tomography images. Med Eng Phys. 2017 Sep;47:105-116. doi: 10.1016/j.medengphy.2017.06.027. Epub 2017 Jul 12. PMID 28711588
- [Background] Li Y, Gutierrez-Chico JL, Holm NR, Yang W, Hebsgaard L, Christiansen EH, Maeng M, Lassen JF, Yan F, Reiber JH, Tu S. Impact of Side Branch Modeling on Computation of Endothelial Shear Stress in Coronary Artery Disease: Coronary Tree Reconstruction by Fusion of 3D Angiography and OCT. J Am Coll Cardiol. 2015 Jul 14;66(2):125-35. doi: 10.1016/j.jacc.2015.05.008. PMID 26160628
- [Background] Torii R, Stettler R, Raber L, Zhang YJ, Karanasos A, Dijkstra J, Patel K, Crake T, Hamshere S, Garcia-Garcia HM, Tenekecioglu E, Ozkor M, Baumbach A, Windecker S, Serruys PW, Regar E, Mathur A, Bourantas CV. Implications of the local hemodynamic forces on the formation and destabilization of neoatherosclerotic lesions. Int J Cardiol. 2018 Dec 1;272:7-12. doi: 10.1016/j.ijcard.2018.06.065. Epub 2018 Jun 19. PMID 30293579
- [Background] Tenekecioglu E, Torii R, Sotomi Y, Collet C, Dijkstra J, Miyazaki Y, Crake T, Su S, Costa R, Chamie D, Liew HB, Santoso T, Onuma Y, Abizaid A, Bourantas CV, Serruys PW. The Effect of Strut Protrusion on Shear Stress Distribution: Hemodynamic Insights From a Prospective Clinical Trial. JACC Cardiovasc Interv. 2017 Sep 11;10(17):1803-1805. doi: 10.1016/j.jcin.2017.06.020. No abstract available. PMID 28882287
- [Background] Torii R, Tenekecioglu E, Katagiri Y, Chichareon P, Sotomi Y, Dijkstra J, Asano T, Modolo R, Takahashi K, Jonker H, van Geuns R, Onuma Y, Pekkan K, Bourantas CV, Serruys PW. The impact of plaque type on strut embedment/protrusion and shear stress distribution in bioresorbable scaffold. Eur Heart J Cardiovasc Imaging. 2020 Apr 1;21(4):454-462. doi: 10.1093/ehjci/jez155. PMID 31215995
- [Background] Papafaklis MI, Bourantas CV, Yonetsu T, Vergallo R, Kotsia A, Nakatani S, Lakkas LS, Athanasiou LS, Naka KK, Fotiadis DI, Feldman CL, Stone PH, Serruys PW, Jang IK, Michalis LK. Anatomically correct three-dimensional coronary artery reconstruction using frequency domain optical coherence tomographic and angiographic data: head-to-head comparison with intravascular ultrasound for endothelial shear stress assessment in humans. EuroIntervention. 2015 Aug;11(4):407-15. doi: 10.4244/EIJY14M06_11. PMID 24974809
- [Background] Papafaklis MI, Bourantas CV, Farooq V, Diletti R, Muramatsu T, Zhang Y, Fotiadis DI, Onuma Y, Garcia Garcia HM, Michalis LK, Serruys PW. In vivo assessment of the three-dimensional haemodynamic micro-environment following drug-eluting bioresorbable vascular scaffold implantation in a human coronary artery: fusion of frequency domain optical coherence tomography and angiography. EuroIntervention. 2013 Nov;9(7):890. doi: 10.4244/EIJV9I7A147. No abstract available. PMID 23856322
- [Background] Bourantas CV, Papafaklis MI, Lakkas L, Sakellarios A, Onuma Y, Zhang YJ, Muramatsu T, Diletti R, Bizopoulos P, Kalatzis F, Naka KK, Fotiadis DI, Wang J, Garcia Garcia HM, Kimura T, Michalis LK, Serruys PW. Fusion of optical coherence tomographic and angiographic data for more accurate evaluation of the endothelial shear stress patterns and neointimal distribution after bioresorbable scaffold implantation: comparison with intravascular ultrasound-derived reconstructions. Int J Cardiovasc Imaging. 2014 Mar;30(3):485-94. doi: 10.1007/s10554-014-0374-3. Epub 2014 Jan 24. PMID 24458955
- [Background] Stone PH, Saito S, Takahashi S, Makita Y, Nakamura S, Kawasaki T, Takahashi A, Katsuki T, Nakamura S, Namiki A, Hirohata A, Matsumura T, Yamazaki S, Yokoi H, Tanaka S, Otsuji S, Yoshimachi F, Honye J, Harwood D, Reitman M, Coskun AU, Papafaklis MI, Feldman CL; PREDICTION Investigators. Prediction of progression of coronary artery disease and clinical outcomes using vascular profiling of endothelial shear stress and arterial plaque characteristics: the PREDICTION Study. Circulation. 2012 Jul 10;126(2):172-81. doi: 10.1161/CIRCULATIONAHA.112.096438. Epub 2012 Jun 21. PMID 22723305
- [Background] Thondapu V, Bourantas CV, Foin N, Jang IK, Serruys PW, Barlis P. Biomechanical stress in coronary atherosclerosis: emerging insights from computational modelling. Eur Heart J. 2017 Jan 7;38(2):81-92. doi: 10.1093/eurheartj/ehv689. PMID 28158723